CLINICAL TRIAL: NCT04905251
Title: Prospective Non Interventional Phase IV Multi-centre Canadian Study on the Effectiveness and Safety of Combination Mifepristone/Misoprostol for Medical Abortion Under 63 Days Gestation
Brief Title: Effectiveness and Safety of Combination Mifepristone/Misoprostol for Medical Abortion
Acronym: MiMAC
Status: Terminated | Type: Observational
Why Stopped: Insufficient Enrollment for Meaningful Analysis/Incomplete or Inconclusive Data Collection. Reaching desired participation numbers of subjects and site was determined to be unfeasible within the two year time period the study was intended to last.
Sponsor: Linepharma International LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: LPI011
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Medical Abortion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Mifepristone-Misoprostol — Non interventional design.

SUMMARY:
National multi-center non interventional study aiming at investigating the effectiveness and safety of the combination mifepristone-misoprostol prescribed in Canada to women for medical termination of pregnancy at or before 63 days gestational age through a multi-center prospective non interventional study design.

DETAILED DESCRIPTION:
Primary Objectives:

* Effectiveness of mifepristone-misoprostol for medical abortion at or prior to 63 days gestational age, defined as complete abortion without further intervention within 14 days of mifepristone administration
* Safety of mifepristone-misoprostol for medical abortion at or prior to 63 days gestational age, defined as the rate of significant Treatment Emergent Adverse Events (TEAE) as a composite outcome of the following events: 1. Hospital Admission; 2. Treatment in Emergency Room; 3. Blood Transfusion; 4. Infection requiring IV Antibiotics, Admission, or Surgical debridement; 5. Death; 6. Ongoing intrauterine pregnancy; 7. Ectopic pregnancy.

Secondary objectives:

* To determine the rate of ongoing pregnancy within 14 days after the administration of mifepristone
* To determine the rate of surgical aspiration performed at the follow-up and time since mifepristone administration
* To determine the reasons for surgical aspiration
* To evaluate the follow-up rate
* To evaluate the delay between the scheduled and actual treatment administration
* To determine the overall safety profile of mifepristone-misoprostol combination
* To evaluate the impact of the demographic characteristics (prescription site, region, gestational age) on effectiveness and safety
* To evaluate the impact of gestational age on effectiveness and safety
* To evaluate the impact of treatment self-administration on effectiveness and safety
* To evaluate the impact of the method and timing of determining gestational age on effectiveness and safety

Study population:

Study performed on a stratified sample of sequential participants (n=3,000) who fulfill trial selection criteria and provide informed consent across a range of clinical practices in Canada (n=30)

ELIGIBILITY:
Inclusion criteria

Women who:

* request elective pregnancy termination in one of the sites participating into the study
* are prescribed mifepristone-misoprostol for this purpose
* provide informed consent to participate in the study.

Exclusion Criteria:

* Participant who is unable to understand or comply with Health Care Professional instructions or medical abortion regimen
* Participant who is unable or unwilling to provide written informed consent.

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — pregnant women
Study Population: Stratified sample of sequential pregnant women requesting medical abortion under 63 days of gestation, who fulfill trial selection criteria and provide informed consent across a range of clinical practices in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2022-02-19 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Effectiveness of mifepristone-misoprostol for medical abortion at or prior to 63 days of gestational age | 14 to 28 days
  Defined as complete abortion without further intervention within 14 days of mifepristone administration.
Safety of mifepristone-misoprostol for medical abortion at or prior to 63 days gestational age | 14 to 28 days
  Defined as the rate of significant Treatment Emergent Adverse Events (TEAE) as a composite outcome of the following events: 1. Hospital Admission; 2. Treatment in Emergency Room; 3. Blood Transfusion; 4. Infection requiring IV Antibiotics, Admission, or Surgical debridement; 5. Death; 6. Ongoing intrauterine pregnancy; 7. Ectopic pregnancy.

SECONDARY OUTCOMES:
Rate of ongoing pregnancy | 14 to 28 days
  Frequency of ongoing pregnancy documented at the first follow-up visit within 14 days after mifepristone administration. The method used to document the completion of abortion and the intervention proposed in case of ongoing pregnancy will also be recorded.
Rate of surgical aspiration | 14-28 days
  Description of the frequency (n and percentage of surgical abortion)
Reasons for surgical aspiration | 14-28 days
  Frequency of the following indications: Ongoing pregnancy, Persistent gestational sac, Retained products of conception, Severe bleeding , Pelvic pain, Suspicion of ectopic pregnancy, others
Delay between the scheduled and actual treatment administration | 14 days
  Measure of the time (in days) between the date scheduled at the initial visit and the actual date of administration of mifepristone.
  Measure of the time (in hour) between the actual administration of misoprostol and the actual administration of mifepristone.
  Description of the rate of mifepristone administration after 63 weeks of gestational age
Overall safety profile of mifepristone-misoprostol combination | 14-28 days
  Frequency of the following:
  * TEAEs /Serious TEAEs (STEAEs) included in the composite criteria,
  * Hysterectomy, Asthma resistant to common drugs, Cardiovascular event, Skin rash, angioedema, anaphylaxis,, Seizure, Suicide,
  * Potential consequences of ongoing pregnancy exposed to mifepristone +/- misoprostol,
  * All other serious adverse events (SAEs) described by System, Organ, Class (SOC) and Preferred Term (PT) ,
  * All other TEAE described by SOC and PT
Impact of the demographic characteristics on effectiveness and safety | 14-28 days
  Comparison of the rates of the primary effectiveness and safety endpoints according to the following stratified parameters:
  * Health Care Professional's site: 1) Abortion Clinic 2) Hospital 3) Private practice 4) Other
  * Type of Health Care Professional: 1) Specialist, 2) General Practitioner, 3) Nurse, 4) Other
  * Participant location : rural vs. urban
  * Geographic area of the prescribing site according to Canadian province
Impact of gestational age on effectiveness and safety | 14-28 days
  Comparison of the rates of the primary effectiveness and safety endpoints according to gestational age at the time of actual mifepristone administration according to the following stratification:
  * ≤ 35 days
  * 36-49 days
  * 50-63 days
  * > 63 days
Impact of treatment self-administration on effectiveness and safety | 14-28 days
  Comparison of the rates of the primary effectiveness and safety endpoints according to the location at which mifepristone is taken:
  * At the study site
  * At home
Impact of the method and timing of determining gestational age on effectiveness and safety | 14-28 days
  Comparison of the rates of the primary effectiveness and safety endpoints according to the fact that ultra-sonography was performed (or not) to confirm gestational age and rule out ectopic pregnancy.
  Description of the mean timing of gestational age determination by ultra-sonography (in weeks of amenorrhea) according to the primary endpoints (existence of complete abortion (yes/no) and of significant treatment emergent adverse event (yes/no)).
Follow-up rate | 28 days
  The follow-up rate will be assessed up to 28 days after mifepristone administration by describing the rate of:
  * Attendance at the in-person follow-up visit between 7 and 14 days after mifepristone administration
  * Attendance at a remote follow-up visit (phone call) up to 28 days after mifepristone administration
  * Loss to follow-up (inability to contact participant up to 28 days following mifepristone administration)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin COSTESCU, MDMS FRCSC, Principal Investigator — McMaster University Medical Centre - Hamilton ON Canada
Locations (6):
- Canada (6):
  - Family Planning Clinic, Moncton City Hospital, Moncton, New Brunswick
  - Centennial Primary Care, Kentville, Nova Scotia
  - Mud Creek Medical, New Minas, Nova Scotia
  - Manitoulin Health Centre, Mindemoya, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Choice in Health Clinic, Toronto, Ontario